CLINICAL TRIAL: NCT03914287
Title: Prospective and Multicenter Study to Assess the Safety and Effectiveness of a Physiotherapy Treatment Through Self-myofascial Release With Foam Roller in Patients With Hemophilic Ankle Arthropathy. A Randomized Clinical Trial.
Brief Title: Self-myofascial Release With Foam Roller in Patients With Hemophilic Ankle Arthropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: He-Foam
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-myofascial release (Experimental): Each session will last approximately 15 minutes, with five physiotherapy sessions taking place over a period of 3 months. The Self-Myofascial release protocol for the lower limbs using a Foam Roller and and Solid Ball Massage, adapted to patients with hemophilic ankle arthropathy will include 11 exercises that must be administered bilaterally. A mobile application will be developed where each patient will be able to observe the exercises to be carried out.
  Interventions: Other: Self-Myofascial release
- Control (No Intervention): Patients included in the control group will not receive any physiotherapy intervention. They will continue with their routine prior to the beginning of the study.

INTERVENTIONS:
Other: Self-Myofascial release — The Self-Myofascial release protocol for the lower limbs using a Foam Roller will include: Self-Myofascial release of the plantar region using and Solid Ball Massage; release of the myofascial components of the back of the leg using a Foam Roller; release of the myofascial components of the anterior part of the leg using a Foam Roller; release of myofascial components of the hamstring region using a Foam Roller; release of the myofascial components of the adductor muscles using a Solid Ball Massage in a sitting position; release of the myofascial components of the abductor muscles using a Foam Roller in lateral decubitus; and release of the myofascial components of the pelvitrochanteric muscles using a Foam Roller in a sitting position.
  Arms: Self-myofascial release

SUMMARY:
Introduction: Hemophilic ankle arthropathy is manifested by degenerative functional alterations (deficit of muscle strength, mobility and proprioception) (intra-articular alterations) and chronic pain. Myofascial release techniques are used to treat soft tissue adhesions, relieve pain and reduce tissue sensitivity.

Design. A randomized clinical trial. Aimed: To evaluate the safety and effectiveness of a protocol by self-myofascial release with Foam Roller applied in patients with hemophilic ankle arthropathy.

Patients: 70 patients with ankle arthropathy will be recruited for inclusion in the study. Patients will be recruited in 5 centers, from different regions of Spain.

Intervention: Each session will last approximately 15 minutes, with five physiotherapy sessions per week for a period of 3 months. Patients will be evaluated at baseline, after the intervention, and after a follow-up period of 3 months. The treatment program includes 11 exercises that must be administered bilaterally. A mobile application will be developed where each patient will be able to observe the exercises to be carried out.

Measuring instruments and study variables: digital goniometer (ankle range of motion); visual analog scale and pressure algometer (joint pain); Haemophilia Joint Health Score (joint status); dynamometer assess (muscle strength); 6-Minute Walking test (functionality of lower limbs); Mobile device (Activity record); Finger-floor test (muscle flexibility). At the same time, the study will allow to determine joint bleeding caused by applied physiotherapy treatment.

Expected results: To demonstrate the safety of this Physiotherapy technique in patients with hemophilia. Likewise, an improvement in ankle pain, functionality and joint motion is expected.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A and B disease.
* Over 18 years.
* Diagnosed with hemophilic arthropathy of the ankle (by clinical assessment with the Hemophilia Joint Health Score).
* On prophylactic or on demand treatment with FVIII / FIX concentrates.

Exclusion Criteria:

* Patients without ambulation ability.
* Patients with inhibitors (antibodies to FVIII or FIX).
* Patients with neurological or cognitive alterations that impede the comprehension of the questionnaires and physical tests.
* Not signed the informed consent document.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline ankle joint pain after treatment and at 3 months | Screening visit, within the first seven days after treatment and after three months follow-up visit
  Visual analogic scale (VAS). This scale will be used to evaluate the perception of joint pain, where ankle joint pain ranges from 0 to 10 points (no pain to maximum perceived pain).

SECONDARY OUTCOMES:
Change from baseline ankle joint pain after treatment and at 3 months | Screening visit, within the first seven days after treatment and after three months follow-up visit
  Pressure algometer. Measuring instrument used to evaluate pressure joint pain. The instrument shall consist of a measuring device attached to a hard rubber tip 1.1 cm in diameter. Its sphere shall be calibrated in kg/cm2 with divisions of 0.1 kg/cm2. The pressure algometry methodology applied was based mainly on the study by Hogeweg. Before taking the measurements, patients will be instructed to say "yes" as soon as pressure exerted by the algometer becomes slightly unpleasant. The pressure algometer shall be kept perpendicular to the surface of the skin with the right hand, stabilizing the axis of the instrument using the thumb and index finger of the left hand. The pressure shall be increased at a uniform rate of approximately 1 kg/cm2 per second. As soon as the subject, according to the instructions, says "yes", the pressure will be stopped and the score will be noted.
Change from baseline lower limb functionality after treatment and at 3 months | Screening visit, within the first seven days after treatment and after three months follow-up visit
  Hemophilia Joint Health Score (HJHS). This measuring instrument will be used to evaluate the joint condition of knees, ankles, and elbows. It includes 8 items (inflammation and its duration, pain, atrophy and muscle strength, crepitus, and reduced flexion and extension) ranging from 0 to 20 points per joint (the higher the score, the greater the joint deterioration).
Change from baseline range of motion of ankle after treatment and at 3 months | Screening visit, within the first seven days after treatment and after three months follow-up visit
  Digital Goniometry Ankle ROM shall be measured using a digital goniometer. The assessment can be made with the patient standing. This measuring instrument allows more accurate measurements than those obtained with a universal plastic goniometer.
Change from baseline muscle strength after treatment and at 3 months | Screening visit, within the first seven days after treatment and after three months follow-up visit
  Dynamometry. The maximum isometric strength of the flexor and extensor muscles of the main joints affected in hemophilia (knees and ankles) will be evaluated on both limbs with a manual dynamometer using a mark test. For this test, the rater needs to keep the dynamometer stationary while the patient exerts maximum force against it.
Change from baseline muscle flexibility after treatment and at 3 months | Screening visit, within the first seven days after treatment and after three months follow-up visit
  Fingertip-to-Floor Test. This test is used to assess the degree of flexibility of the posterior muscles of the lower limbs. This value is calculated as the distance between the fingertip and the floor when maximum hip flexion with knee extension is performed.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Real Fundación Victoria Eugenia
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merono-Gallut AJ, Cuesta-Barriuso R, Perez-Llanes R, Donoso-Ubeda E, Lopez-Pina JA. Self-Myofascial Release Intervention and Mobile App in Patients With Hemophilic Ankle Arthropathy: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Jul 31;9(7):e15612. doi: 10.2196/15612. PMID 32734929